CLINICAL TRIAL: NCT04330209
Title: Comparing a Low-GI Nutrigenetic and Ketogenic Diet for Weight Loss With 18 Month Follow-up
Acronym: LOWGI_GENE
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Keith Anthony Grimaldi, Honorary Research Fellow, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: LOWGI_GENE
Record Dates: First submitted 2020-03-27; First posted 2020-04-01 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Weight Loss; Glucose, High Blood; LDL Hyperlipoproteinemia; HDL; Triglycerides High
Keywords: Glycaemic index; nutrigenetics; weight loss; ketogenic; nutrigenomics
MeSH Terms: conditions — Weight Loss; Hypertriglyceridemia | interventions — Diet, Reducing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — buccal swab for DNA, venous blood for cholesterol & glucose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LowGI/nutrigenetic: 114 overweight (n=1) and obese (n=113) subjects (M = 55, F = 59, age 24-56y, all of Romanian heritage and similar socio-economic status), who were patients at a weight management clinic (Bucharest, Romania), gave written informed consent for their weight loss data to be prospectively analysed for this study.
  Upon enrolment at the weight management clinic, the subjects self-selected either a ketogenic diet or a low-GI nutrigenetic diet. 61 subjects (34 female; age 42.0 ± 6.7y) selected the low-GI nutrigenetic diet plan.
  Interventions: Other: weight loss diets
- Ketogenic: As above + Fifty-three subjects (25 female; age 43.0 ± 7.2y) selected the ketogenic diet plan
  Interventions: Other: weight loss diets

INTERVENTIONS:
Other: weight loss diets — The ketogenic diet group were instructed to consume <35g of carbohydrates per day, and <10% of total calories were from saturated fats. Daily protein intake was set at 1.2g/kg bodyweight for females, and 1.5g/kg bodyweight for males. The low-GI nutrigenetic diet group had individualised dietary instructions based on their genetic results

SUMMARY:
The investigators followed a convenience sample of 114 overweight and obese subjects from a weight loss clinic who followed a 24-week dietary intervention. The subjects self-selected whether to follow a standardized ketogenic diet (n=53), or a personalised low-glycemic index (GI) diet utilising information from 28 single nucleotide polymorphisms (n=61). After the 24-week study period, the subjects were monitored for an additional 18 months.

DETAILED DESCRIPTION:
In the present study, the investigators followed patients in a clinic who self-selected either a ketogenic diet with no nutrigenetic modification, or a low glycemic index (GI) based diet with nutrigenetic modifications. The addition of nutrigenetic advice was not designed nor proposed to patients as a weight loss diet, nor to predict either disease risk or obesity risk; the aim was simply to optimize the nutrient content of an individual's daily food intake, based on current understanding of an individual's genetic profile. The aim of this study, therefore, was to compare the performance of the well-known, and generally the most effective in the short-term [25], ketogenic diet to a low-GI nutrigenetic diet. A ketogenic diet has also shown to have long-term (12 months) effectiveness for weight loss [26], although the effects of the diet over a longer time period than this are currently unclear.

114 overweight (n=1) and obese (n=113) subjects (M = 55, F = 59, age 24-56y, all of Romanian heritage and similar socio-economic status), who were patients at a weight management clinic (Bucharest, Romania), gave written informed consent for their weight loss data to be prospectively analysed for this study. All patient data were handled according to the Romanian Code of Medical Deontology and in accordance with the Helsinki Agreement. Approval was given by the Ethics Committee of the University and Pharmacy, Cluj Napoca, Romania (registration number 444). Upon enrolment at the weight management clinic, the subjects self-selected either a ketogenic diet or a low-GI nutrigenetic diet. A ketogenic diet was utilised as the comparison diet due to its reported efficacy in the treatment of obesity [26]. Fifty-three subjects (25 female; age 43.0 ± 7.2y) selected the ketogenic diet plan, and 61 subjects (34 female; age 42.0 ± 6.7y) selected the low-GI nutrigenetic diet plan. Subjects in the low-GI nutrigenetic diet group underwent DNA testing (NutriGENE by Eurogenetica Ltd/DNAfit, UK) for 28 Single Nucleotide Polymorphisms (SNPs) in 22 genes with good evidence of gene-diet/lifestyle interactions [table 1]. Overall participation in both diet groups cost a similar amount, comprised of approximately €300 for the genetic test along with 1-month diet plan, initial evaluation, body composition, and medical history for the nutrigenetic group, and €280 for the ketogenic group, providing Ketostix and the same evaluations. Further visits through the 24-week program the overall cost per patient was approximately €800. After 24 weeks diet follow up visits had no further cost.

After the 24-week study period, the subjects were monitored for an additional 18 months.

At the study onset, patients were not type 1 or type 2 diabetics, although many were hyperglycemic, which is a common issue in obese subjects. Any patients with records of any other disease were excluded prior to commencing the dietary intervention. The patients, apart from obesity, were otherwise "healthy".

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI ≥30)
* Age ≥ 18 years
* Male or female
* Smoking or not smoking

Exclusion Criteria:

* Type 1 diabetes
* Type 2 diabetes
* Any other disease

Ages: 24 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 114 overweight (n=1) and obese (n=113) subjects (M = 55, F = 59, age 24-56y, all of Romanian heritage and similar socio-economic status
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Weight loss - kg and BMI | 6 months
  Weight loss after 6 months diet
Weight loss - kg and BMI | 18 months
  After 18-months follow up on normal nutrition

SECONDARY OUTCOMES:
Blood glucose | 6 months
  Levels of blood glucose
Blood glucose | 18 months
  Levels of blood glucose
Cholesterol | 6 months
  Levels of LDL and LDL
Cholesterol | 18 months
  Levels of LDL and LDL
Triglycerides | 6 months
  Levels of blood triglycerides
Triglycerides | 18 months
  Levels of blood triglycerides

IPD SHARING:
Plan to Share IPD: Undecided
genetic, weight, gender, age, blood biomarker data

REFERENCES:
- [Derived] Vranceanu M, Pickering C, Filip L, Pralea IE, Sundaram S, Al-Saleh A, Popa DS, Grimaldi KA. A comparison of a ketogenic diet with a LowGI/nutrigenetic diet over 6 months for weight loss and 18-month follow-up. BMC Nutr. 2020 Sep 24;6:53. doi: 10.1186/s40795-020-00370-7. eCollection 2020. PMID 32983551